CLINICAL TRIAL: NCT02311582
Title: A Phase I/II Study Testing the Safety, Toxicities, and Efficacy of MK-3475 in Combination With MRI-guided Laser Ablation in Recurrent Malignant Gliomas
Brief Title: MK-3475 in Combination With MRI-guided Laser Ablation in Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201501072
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: As of Amendment 12, patients enrolled in the phase II portion of this trial will no longer be randomized. These patients will undergo MLA followed by MK-3475 treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (5):
- Phase I: MK-3475 + MLA Dose Level 1 (Experimental): MK-3475 will be given at 100 mg intravenously (IV) every 3 weeks starting no more than 1 week after MLA until progression or unacceptable toxicity.
  Interventions: Biological: MK-3475; Device: MRI-guided laser ablation
- Phase I: MK-3475 + MLA Dose Level 2 (Experimental): MK-3475 will be given at 150 mg intravenously (IV) every 3 weeks starting no more than 1 week after MLA until progression or unacceptable toxicity.
  Interventions: Biological: MK-3475; Device: MRI-guided laser ablation
- Phase I: MK-3475 + MLA Dose Level 3 (Experimental): MK-3475 will be given at 200 mg intravenously (IV) every 3 weeks starting no more than 1 week after MLA until progression or unacceptable toxicity.
  Interventions: Biological: MK-3475; Device: MRI-guided laser ablation
- Phase II: MK-3475 + MLA (Experimental): MK-3475 will be given at 200 mg intravenously (IV) every 3 weeks no more than 1 week after MLA, or no more than 1 week after biopsy (if no surgical debulking). This dose was determined in the Phase I portion of the trial.
  Interventions: Biological: MK-3475; Device: MRI-guided laser ablation
- Phase II: MK-3475 Only (Experimental): MK-3475 will be given at 200 mg intravenously (IV) every 3 weeks beginning 3 weeks after surgical debulking or no more than 1 week after biopsy (if no surgical debulking). This dose was determined in the Phase I portion of the trial.
  Interventions: Biological: MK-3475

INTERVENTIONS:
Biological: MK-3475 — Patients currently on pembrolizumab beyond the 2 year/35 cycle limit at the time of the approval of Amendment 13 (approved 07/28/2021) may continue to receive pembrolizumab unless there is progression, toxicity or agreement by the patient and PI to come off therapy. Participants who discontinue pembrolizumab after receiving 35 doses are eligible for retreatment with pembrolizumab if they progress during follow-up provided they meet the requirements. Participants may receive an additional 17 cycles (12 months) of pembrolizumab during the Second Course Phase (Retreatment).
  Other Names: Pembrolizumab; Keytruda
Device: MRI-guided laser ablation — MLA is a minimally invasive laser surgery, which employs a small incision in the scalp and skull, through which a thin laser probe is inserted and guided by MR imaging to the core of the tumor mass where it delivers hyperthermic ablation from the core to the rim.
  Other Names: MLA; NeuroBlate; AutoLITT
  Arms: Phase I: MK-3475 + MLA Dose Level 1; Phase I: MK-3475 + MLA Dose Level 2; Phase I: MK-3475 + MLA Dose Level 3; Phase II: MK-3475 + MLA

SUMMARY:
The blood brain barrier (BBB) is a major obstacle to drug delivery in the treatment of malignant brain tumors including glioblastoma multiforme (GBM). MRI-guided laser ablation (MLA) has been noted to disrupt peritumoral the blood brain barrier (BBB), which may then lead to increased access of new tumor antigens to the lymphovascular system and vice versa of immune effector cells to the tumor for effective activation of the immune system, and tumor infiltration, respectively. Therefore, the combination of MK-3475 and MLA as proposed in this protocol is hypothesized to create a therapeutic combinatorial effect in which MLA increases material access to promote immune activation and then MK-3475 maximizes these tumor-specific immune reactions to impart effective tumor control.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Histologically confirmed grade III or IV malignant glioma.
* Phase II: Histologically confirmed grade IV malignant glioma (GBM).

  *Note: GBM variants and suspected secondary GBM are allowed for both phase I and phase II.
* Unequivocal evidence of tumor progression as documented by biopsy or brain MRI scan per RANO criteria.
* There must be an interval of at least 12 weeks from the completion of standard front-line therapy to study registration unless there is unequivocal evidence for tumor recurrence per RANO criteria. When the interval is less than 12 weeks, the use of perfusion imaging and/or PET scan is allowed to differentiate between unequivocal evidence of tumor recurrence and pseudoprogression. Standard front-line therapy is as described below:

  * For grade IV malignant gliomas (GBM): Standard front line therapy for newly diagnosed GBM must include maximal feasible surgical resection (biopsy alone allowed), radiotherapy, and temozolomide chemotherapy. If the tumor was initially diagnosed as either a grade II or III tumor and now has recurred or progressed as a grade IV GBM, it will be considered a secondary recurrent grade IV GBM and will be eligible for this study as long as prior treatment included maximal feasible surgical resection (biopsy alone allowed), radiotherapy, and temozolomide chemotherapy.
  * For grade III malignant gliomas with 1p 19q codeletions: Standard front line therapy for newly diagnosed grade III malignant gliomas must include maximal feasible surgical resection (biopsy alone allowed), radiotherapy, and chemotherapy (PCV or temozolomide). If the patient did not receive any or all components of the standard front line therapy as detailed above for newly diagnosed grade III gliomas and the tumor then recurred or progressed, s/he must first receive at least one prior standard therapy or any appropriate combination of the components of standard therapy as detailed above and must experience further recurrence or progression before s/he is deemed eligible for this study. If the tumor was initially diagnosed as a grade II glioma with 1p 19q codeletions and now has recurred or progressed as a grade III tumor, it will be considered a secondary recurrent grade III glioma with 1p 19q codeletions and will be eligible for this study as long as prior treatment included maximal feasible surgical resection (biopsy alone allowed), radiotherapy, and chemotherapy (PCV or temozolomide).
  * For grade III malignant gliomas without 1p 19q codeletions: Standard front-line therapy for newly diagnosed grade III malignant gliomas must include maximal feasible surgical resection (biopsy alone allowed), radiotherapy, and temozolomide chemotherapy. If the tumor was initially diagnosed as a grade II glioma without 1p 19q codeletions and now has recurred or progressed as a grade III tumor, it will be considered a secondary recurrent grade III glioma without 1p 19q codeletions and will be eligible for this study as long as prior treatment included maximal feasible surgical resection (biopsy alone allowed), radiotherapy, and temozolomide chemotherapy.
* Candidate for MLA based on the size, location, and shape of the recurrent tumor as determined by the performing neurosurgeon. Surgical resection/debulking prior to MLA is allowed per standard of care but is not required; if the patient undergoes resection or debulking, it must have occurred at least 3 weeks prior to the first dose of MK-3475. For Phase II: if surgical resection/debulking prior to MLA is not indicated, a biopsy of the tumor will be done at the same time of MLA to obtain tumor tissue for both diagnostic purposes and immune monitoring.
* Patients who have undergone a resection for recurrence will be eligible. In those who have undergone a gross total resection, the MLA will be directed at treating a peritumoral margin of 0.5-1cm surrounding the resection cavity to disrupt the BBB and potentially increase access of MK-3475 to the peritumoral infiltrating glioma cells.
* At least 18 years of age.
* Karnofsky ≥ 60%
* Normal bone marrow and organ function as defined below:

  * ANC ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
  * Serum creatinine ≤ 1.5 x IULN OR creatinine clearance by Cockcroft-Gault ≥ 60 mL/min for patients with serum creatinine > 1.5 x IULN
  * Serum total bilirubin ≤ 1.5 x IULN OR direct bilirubin ≤ IULN for patients with total bilirubin > 1.5 x IULN
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 x IULN (or ≤ 5 x IULN for patients with liver metastases)
  * INR or PT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * aPTT ≤ 1.5 x IULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Sexually active women of childbearing potential and men must agree to use contraception (as described in the protocol) prior to study entry, for the duration of study participation, and for 120 days after last dose of MK-3475. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patients with the ability to understand and willingness to sign an IRB approved written informed consent document will be enrolled into the trial. However, should a patient lose their ability to consent while participating in this study and s/he is still receiving clinical benefit from participation, s/he may continue on study with the consent of a Legally Authorized Representative.

Exclusion Criteria:

* Prior treatment with any anti-angiogenic agent (including bevacizumab).
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Prior treatment with a monoclonal antibody within 4 weeks prior to the first dose of MK-3475 or has not recovered (i.e. ≤ grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first dose of MK-3475 or has not recovered (i.e. ≤ grade 1 or at baseline) from adverse events due to a previously administered agent.

  * Note: patients with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study.
  * Note: if a patient underwent major surgery, s/he must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Candidates for curative resection or urgent surgical procedure(s) needed.
* Presence of infratentorial lesions, brainstem lesions, or lesions that are less than 5 mm from the hyophysis or cranial nerves.
* Multifocal gliomas that are bilateral. Patients with unilateral multifocal gliomas may be eligible if their multifocal disease can be treated effectively and safely in a single MLA procedure.
* Presence of leptomeningeal metastases.
* Recent (within 8 weeks) history of CNS hemorrhage unless the hemorrhage is located within the tumor that will be removed en total during surgical debulking or ablated during MLA.
* Requires therapeutic doses of anticoagulants unless anticoagulation can be safely discontinued before surgery per standard practice (e.g. first DVD for which anticoagulation has been at least 3 months and repeat imaging demonstrates resolution of DVT) or an IVC filter can be used in place of anticoagulation. Subjects are permitted to resume anticoagulation following surgery per discretion of treating physician and/or site SOPs
* Received prior local therapy (stereotactic radiosurgery, brachytherapy, or carmustine wafers) to the proposed area of MLA treatment.
* Received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of MK-3475. Administration of killed vaccines is allowed.
* Currently receiving any other investigational agents or has participated in a study of an investigational agent or using an investigational device within 3 weeks of the first dose of MK-3475.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-3475 or other agents used in the study.
* Dexamethasone > 4 mg daily at the time of registration
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment (with the exception of daily dexamethasone ≤ 4 mg).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
* Has an active autoimmune disease requiring systemic treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or current pneumonitis/interstitial lung disease.
* Pregnant and/or breastfeeding. Patient must have a negative serum or urine pregnancy test within 72 hours of study entry.
* Known history of hepatitis B (e.g.,defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (e.g.,defined as HCV RNA [qualitative] is detected) infection.
* Known history of active TB (bacillus tuberculosis).
* Known history of HIV (HIV 1/2 antibodies).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-08-05 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milan G Chheda, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hwang H, Huang J, Khaddour K, Butt OH, Ansstas G, Chen J, Katumba RG, Kim AH, Leuthardt EC, Campian JL. Prolonged response of recurrent IDH-wild-type glioblastoma to laser interstitial thermal therapy with pembrolizumab. CNS Oncol. 2022 Mar 1;11(1):CNS81. doi: 10.2217/cns-2021-0013. Epub 2022 Jan 19. PMID 35043686
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase I: MK-3475 + MLA Dose Level 1 | Phase I: MK-3475 + MLA Dose Level 2 | Phase I: MK-3475 + MLA Dose Level 3 | Phase II: MK-3475 + MLA | Phase II: MK-3475 Only
Started | 3 | 3 | 3 | 36 | 10
Completed | 3 | 3 | 3 | 30 | 6
Not Completed | 0 | 0 | 0 | 6 | 4
Not completed — Was enrolled but did not receive any MK-3475 treatment | 0 | 0 | 0 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: MK-3475 + MLA Dose Level 1 | Phase I: MK-3475 + MLA Dose Level 2 | Phase I: MK-3475 + MLA Dose Level 3 | Phase II: MK-3475 + MLA | Phase II: MK-3475 Only | Total
Number analyzed (Participants) | 3 | 3 | 3 | 36 | 10 | 55
Age, Continuous [Median (Full Range); unit: years] | 57 [57 to 62] | 41 [37 to 49] | 67 [49 to 72] | 60 [33 to 80] | 56.5 [46 to 68] | 57 [33 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 19 | 7 | 31
  Male | 1 | 2 | 1 | 17 | 3 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 3 | 36 | 10 | 54
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 3 | 3 | 34 | 10 | 53
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 36 | 10 | 55

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of MK-3475 When Combined With MLA - Phase I Only
Description: The MTD is defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experienced dose-limiting toxicity during the first cycle. Dose escalations will proceed until the MTD has been reached, or failing that, 200 mg of MK-3475 every 3 weeks will be considered the MTD.
Time Frame: Completion of Cycle 1 (each cycle is 3 weeks)
Measure: Number; unit: mg
Groups:
- Phase I: MK-3475 + MLA: MK-3475 will be given at the assigned dose intravenously (IV) every 3 weeks starting no more than 1 week after MLA until progression or unacceptable toxicity.
Arm/Group | Phase I: MK-3475 + MLA
Number analyzed (Participants) | 9
mg | 200

2. Primary Outcome: Progression-free Survival (PFS) - Phase II Only
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Time Frame: Through completion of follow-up (median length of follow-up 338 days, full range 43-2468 days).
Population: Participants are evaluable for this outcome measure if they were treated in the Phase II portion of the trial (includes Phase II MK-3475 + MLA and Phase II MK-3475 Only) and at the MTD in Phase I (MK-3475 + MLA Dose Level 3). The Phase I MTD is included with the Phase II MK-3475 + MLA arm since the patients received the same dosing of treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase I MTD + Phase II: MK-3475 + MLA: MK-3475 will be given at 200 mg intravenously (IV) every 3 weeks no more than 1 week after MLA, or no more than 1 week after biopsy (if no surgical debulking). This dose was determined in the Phase I portion of the trial.
Arm/Group | Phase I MTD + Phase II: MK-3475 + MLA | Phase II: MK-3475 Only
Number analyzed (Participants) | 33 | 6
months | 5.3 [3.4 to 12.4] | 2.1 [0.99 to NA] — The upper 95% confidence interval is not available as there is an insufficient number of participants with events.

3. Secondary Outcome: Toxicity Profile of MK-3475 in Combination With MLA - Phase I Only
Description: * The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting
  * The only toxicities that will not be collected are those that are clearly related to MLA and/or surgery AND ALSO not related to MK-3475
  * Adverse events will be tracked from start of treatment through 30 days following the last day of study treatment. Serious adverse events will be tracked for 90 days following the last dose of study treatment.
Time Frame: Through 90 days after completion of treatment (up to 168 weeks)
Population: Participants in Phase II were not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: MK-3475 + MLA Dose Level 1 | Phase I: MK-3475 + MLA Dose Level 2 | Phase I: MK-3475 + MLA Dose Level 3 | Phase II: MK-3475 + MLA | Phase II: MK-3475 Only
Number analyzed (Participants) | 3 | 3 | 3 | 0 | 0
Participants
  Grade 1/2 anemia | 1 | 1 | 1 |  |
  Grade 3/4/5 lactic acidosis | 0 | 0 | 1 |  |
  Grade 3/4/5 leukocytosis | 0 | 0 | 1 |  |
  Grade 1/2 tachycardia | 0 | 1 | 0 |  |
  Grade 1/2 blurred vision | 1 | 0 | 1 |  |
  Grade 1/2 drooping eyes | 0 | 0 | 1 |  |
  Grade 1/2 floaters | 1 | 0 | 0 |  |
  Grade 1/2 glaucoma | 0 | 0 | 1 |  |
  Grade 1/2 pressure around eyes | 0 | 0 | 1 |  |
  Grade 1/2 right visual field cut | 0 | 0 | 1 |  |
  Grade 1/2 swollen eyes | 0 | 0 | 1 |  |
  Grade 3/4/5 abdominal pain | 0 | 1 | 0 |  |
  Grade 1/2 diarrhea | 0 | 0 | 1 |  |
  Grade 3/4/5 diarrhea | 0 | 3 | 0 |  |
  Grade 1/2 dysphagia | 1 | 0 | 0 |  |
  Grade 1/2 nausea | 1 | 0 | 0 |  |
  Grade 1/2 oral pain | 0 | 0 | 1 |  |
  Grade 1/2 rectal hemorrhage | 0 | 0 | 1 |  |
  Grade 1/2 vomiting | 1 | 0 | 0 |  |
  Grade 1/2 edema face | 0 | 1 | 1 |  |
  Grade 1/2 edema limbs | 0 | 0 | 1 |  |
  Grade 1/2 fatigue | 1 | 2 | 1 |  |
  Grade 1/2 fever | 0 | 1 | 0 |  |
  Grade 1/2 infusion related reaction | 0 | 1 | 0 |  |
  Grade 1/2 pain | 0 | 0 | 1 |  |
  Grade 3/4/5 appendicitis | 1 | 0 | 0 |  |
  Grade 1/2 bronchial infection | 0 | 0 | 1 |  |
  Grade 3/4/5 cellulitis | 0 | 0 | 1 |  |
  Grade 1/2 cold | 0 | 1 | 0 |  |
  Grade 1/2 pneumonia | 1 | 0 | 0 |  |
  Grade 3/4/5 sepsis | 0 | 0 | 1 |  |
  Grade 1/2 urinary tract infection | 1 | 0 | 0 |  |
  Grade 3/4/5 urinary tract infection | 0 | 1 | 0 |  |
  Grade 1/2 bruising | 0 | 1 | 1 |  |
  Grade 1/2 fall | 0 | 1 | 2 |  |
  Grade 3/4/5 fracture | 0 | 0 | 1 |  |
  Grade 1/2 wound from fall | 0 | 0 | 1 |  |
  Grade 1/2 alanine aminotransferase increased | 0 | 1 | 0 |  |
  Grade 1/2 alkaline phosphatase increased | 0 | 1 | 0 |  |
  Grade 1/2 blood bilirubin increased | 0 | 0 | 1 |  |
  Grade 1/2 creatinine increased | 1 | 0 | 1 |  |
  Grade 1/2 lymphocyte count decreased | 0 | 3 | 2 |  |
  Grade 1/2 platelet count decreased | 2 | 0 | 1 |  |
  Grade 1/2 weight loss | 0 | 0 | 1 |  |
  Grade 1/2 white blood cell decreased | 2 | 1 | 0 |  |
  Grade 1/2 hyperglycemia | 3 | 1 | 0 |  |
  Grade 3/4/5 hyperglycemia | 0 | 0 | 1 |  |
  Grade 1/2 hyperkalemia | 0 | 0 | 1 |  |
  Grade 1/2 hypernatremia | 0 | 0 | 1 |  |
  Grade 1/2 hypoalbuminemia | 0 | 1 | 0 |  |
  Grade 1/2 hyponatremia | 0 | 0 | 1 |  |
  Grade 1/2 arthritis | 0 | 0 | 1 |  |
  Grade 1/2 back pain | 0 | 1 | 1 |  |
  Grade 1/2 chest wall pain | 0 | 1 | 0 |  |
  Grade 1/2 dystonia | 0 | 1 | 0 |  |
  Grade 1/2 generalized muscle weakness | 0 | 0 | 1 |  |
  Grade 1/2 joint effusion | 1 | 0 | 0 |  |
  Grade 1/2 muscle weakness - left sided | 1 | 1 | 0 |  |
  Grade 1/2 muscle weakness - right sided | 0 | 1 | 0 |  |
  Grade 3/4/5 muscle weakness - right sided | 0 | 0 | 1 |  |
  Grade 1/2 muscle weakness - upper limb | 0 | 0 | 1 |  |
  Grade 1/2 pain in extremity | 0 | 1 | 0 |  |
  Grade 3/4/5 altered mental status | 0 | 1 | 0 |  |
  Grade 1/2 cognitive disturbance | 1 | 0 | 0 |  |
  Grade 1/2 dizziness | 1 | 1 | 1 |  |
  Grade 1/2 edema cerebral | 0 | 1 | 0 |  |
  Grade 1/2 expressive aphasia | 0 | 1 | 0 |  |
  Grade 1/2 headache | 1 | 1 | 2 |  |
  Grade 3/4/5 intracranial hemorrhage | 0 | 0 | 1 |  |
  Grade 1/2 lethargy | 1 | 1 | 0 |  |
  Grade 1/2 lightheadedness | 1 | 0 | 0 |  |
  Grade 1/2 memory impairment | 0 | 0 | 1 |  |
  Grade 3/4/5 peripheral motor neuropathy | 0 | 1 | 0 |  |
  Grade 1/2 reading comprehension difficulty | 1 | 0 | 0 |  |
  Grade 3/4/5 seizure | 1 | 1 | 0 |  |
  Grade 3/4/5 speech aphasia | 0 | 0 | 1 |  |
  Grade 1/2 word-finding difficulty | 1 | 0 | 0 |  |
  Grade 1/2 agitation | 0 | 1 | 0 |  |
  Grade 1/2 anxiety | 1 | 0 | 1 |  |
  Grade 1/2 confusion | 0 | 0 | 1 |  |
  Grade 1/2 insomnia | 0 | 1 | 0 |  |
  Grade 1/2 hematuria | 0 | 0 | 2 |  |
  Grade 1/2 urinary incontinence | 0 | 0 | 1 |  |
  Grade 1/2 cough | 1 | 1 | 1 |  |
  Grade 1/2 dyspnea | 1 | 0 | 1 |  |
  Grade 1/2 nasal congestion | 0 | 1 | 0 |  |
  Grade 1/2 dry skin | 0 | 1 | 1 |  |
  Grade 1/2 hyperhidrosis | 0 | 0 | 1 |  |
  Grade 3/4/5 rash | 0 | 1 | 0 |  |
  Grade 3/4/5 skin ulceration | 0 | 1 | 0 |  |
  Grade 3/4/5 planned left craniectomy | 0 | 0 | 1 |  |
  Grade 1/2 hot flashes | 1 | 0 | 1 |  |
  Grade 1/2 hypertension | 0 | 0 | 1 |  |
  Grade 3/4/5 hypotension | 1 | 0 | 0 |  |
  Grade 3/4/5 pulmonary embolism | 0 | 1 | 0 |  |

4. Secondary Outcome: Overall Survival (OS) - Phase II Only
Description: OS is defined as the duration of time from start of treatment to time of death.
Time Frame: Through completion of follow-up (median length of follow-up 338 days, full range 43-2468 days).
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I MTD + Phase II: MK-3475 + MLA | Phase II: MK-3475 Only
Number analyzed (Participants) | 33 | 6
months | 11.8 [8.9 to 27.7] | 5.2 [1.7 to NA] — The upper 95% confidence interval is not available as there is an insufficient number of participants with events.

5. Secondary Outcome: Anti-glioma Immune Response Before and After MK-3475 With MLA - Phase II Only
Time Frame: Up to 26 months
Population: Patients underwent pre-LITT surgery or biopsy concurrent with LITT with resulting tissue (no minimum tissue volume requirement) first determining eligibility & any remaining tissue made available for the analyses listed in the secondary outcome measures. In practice, concurrent local biopsy was heavily favored over two stage surgeries for study participants. Biopsy provided comparatively smaller volumes of tissue &, unfortunately ended up not providing adequate tissue for this analysis.
Arm/Group | Phase I: MK-3475 + MLA Dose Level 1 | Phase I: MK-3475 + MLA Dose Level 2 | Phase I: MK-3475 + MLA Dose Level 3 | Phase II: MK-3475 + MLA | Phase II: MK-3475 Only
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Correlate Intratumoral Expression of PD-L1 and the Frequency of Glioma Cell-specific Cytotoxic T Cells With PFS - Phase II Only
Time Frame: 6 months
Population: as for outcome 5
Arm/Group | Phase I: MK-3475 + MLA Dose Level 1 | Phase I: MK-3475 + MLA Dose Level 2 | Phase I: MK-3475 + MLA Dose Level 3 | Phase II: MK-3475 + MLA | Phase II: MK-3475 Only
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Correlate Intratumoral Expression of PD-L1 and the Frequency of Glioma Cell-specific Cytotoxic T Cells With OS - Phase II Only
Time Frame: Up to 2 years after completion of treatment (estimated to be up to 272 weeks)
Population: as for outcome 5
Arm/Group | Phase I: MK-3475 + MLA Dose Level 1 | Phase I: MK-3475 + MLA Dose Level 2 | Phase I: MK-3475 + MLA Dose Level 3 | Phase II: MK-3475 + MLA | Phase II: MK-3475 Only
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Identify PD-1-dependent Biomarkers in Glioma Cell-specific T Cells That Negatively Correlate With the Frequency of Glioma Cell-specific Cytotoxic T Cells and PFS - Phase II Only
Time Frame: Up to 2 years after completion of treatment (estimated to be up to 272 weeks)
Population: as for outcome 5
Arm/Group | Phase I: MK-3475 + MLA Dose Level 1 | Phase I: MK-3475 + MLA Dose Level 2 | Phase I: MK-3475 + MLA Dose Level 3 | Phase II: MK-3475 + MLA | Phase II: MK-3475 Only
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Identify PD-1-dependent Biomarkers in Glioma Cell-specific T Cells That Negatively Correlate With the Frequency of Glioma Cell-specific Cytotoxic T Cells and OS - Phase II Only
Time Frame: Up to 2 years after completion of treatment (estimated to be up to 272 weeks)
Population: as for outcome 5
Arm/Group | Phase I: MK-3475 + MLA Dose Level 1 | Phase I: MK-3475 + MLA Dose Level 2 | Phase I: MK-3475 + MLA Dose Level 3 | Phase II: MK-3475 + MLA | Phase II: MK-3475 Only
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were followed from start of MK-3475 through 30 days following the last day of treatment (median length of follow-up 152 days, full range 43-1778 days). Serious adverse events were followed from start of MK-3475 through 90 days following the last day of treatment (median length of follow-up 212 days, full range 43-1838 days). All-cause mortality was followed from start of MK-3475 through completion of follow-up (median length of follow-up 338 days, full range 43-2468 days).
Arm/Group | Phase I: MK-3475 + MLA Dose Level 1 | Phase I: MK-3475 + MLA Dose Level 2 | Phase I: MK-3475 + MLA Dose Level 3 | Phase II: MK-3475 + MLA | Phase II: MK-3475 Only
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 1/3 | 26/30 | 5/6
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 2/3 | 15/30 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 30/30 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: MK-3475 + MLA Dose Level 1 (N=3) | Phase I: MK-3475 + MLA Dose Level 2 (N=3) | Phase I: MK-3475 + MLA Dose Level 3 (N=3) | Phase II: MK-3475 + MLA (N=30) | Phase II: MK-3475 Only (N=6)
Lactic acidosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Fever (General disorders) | 0 | 1 | 0 | 0 | 0
Lethargy (General disorders) | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes zoster infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Prolonged hospitalization following MLA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Recurrent glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral edema (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Left-sided weakness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Right-sided weakness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 2 | 0 | 4 | 0
Speech aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Altered mental status (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Planned left craniectomy (Surgical and medical procedures) | 0 | 0 | 1 | 1 | 0
Planned post-progression Monteris Laser Ablation procedure (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Planned post-progression surgical resection (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Ventriculoperitoneal shunt placement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: MK-3475 + MLA Dose Level 1 (N=3) | Phase I: MK-3475 + MLA Dose Level 2 (N=3) | Phase I: MK-3475 + MLA Dose Level 3 (N=3) | Phase II: MK-3475 + MLA (N=30) | Phase II: MK-3475 Only (N=6)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 6 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Balance issues (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 5 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 1 | 0 | 1 | 3 | 0
Drooping eyes (Eye disorders) | 0 | 0 | 1 | 0 | 0
Floaters (Eye disorders) | 1 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0
Pressure around eyes (Eye disorders) | 0 | 0 | 1 | 0 | 0
Right eye visual disturbance (Eye disorders) | 0 | 0 | 0 | 0 | 1
Right peripheral field deficit (Eye disorders) | 0 | 0 | 0 | 0 | 1
Right visual field cut (Eye disorders) | 0 | 0 | 1 | 0 | 0
Swollen eyes (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision changes (Eye disorders) | 0 | 0 | 0 | 2 | 0
Worsening right visual field cut (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 3 | 1 | 8 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Gastroesophageal reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Chills (General disorders) | 0 | 0 | 0 | 1 | 0
Edema (General disorders) | 0 | 0 | 0 | 0 | 1
Edema face (General disorders) | 0 | 1 | 1 | 3 | 1
Edema limbs (General disorders) | 0 | 0 | 1 | 4 | 0
Fatigue (General disorders) | 1 | 2 | 1 | 16 | 3
Fever (General disorders) | 0 | 0 | 0 | 2 | 0
Fluid collection from elbow (General disorders) | 0 | 0 | 0 | 1 | 0
Infusion related reaction (General disorders) | 0 | 1 | 0 | 0 | 0
Left shoulder pain (General disorders) | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 6 | 1
Bronchial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
COVID-19 infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cold (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Mucosal - Thrush (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 5 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post-operative aphasia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound - finger laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound from fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Activated thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 5 | 2
Alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1 | 0
Creatinine increased (Investigations) | 1 | 0 | 1 | 2 | 0
Hemoglobin increased (Investigations) | 0 | 0 | 0 | 1 | 0
INR increased (Investigations) | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 3 | 2 | 22 | 5
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2 | 0
Platelet count decreased (Investigations) | 2 | 0 | 1 | 4 | 3
Weight gain (Investigations) | 0 | 0 | 0 | 6 | 1
Weight loss (Investigations) | 0 | 0 | 1 | 2 | 0
White blood cell decreased (Investigations) | 2 | 1 | 0 | 5 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 7 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 4 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Dystonia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 4 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Upper limb muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0 | 5 | 0
Concentration impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 5 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 0 | 0 | 7 | 1
Edema cerebral (Nervous system disorders) | 0 | 1 | 0 | 2 | 0
Expressive aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Gait disturbance (Nervous system disorders) | 0 | 0 | 0 | 3 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 12 | 5
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Irritability (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lightheadedness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 3 | 2
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 5 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Pseduomeningocele (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Reading comprehension difficulty (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Speech and coordination (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 4 | 0
Word-finding difficulty (Nervous system disorders) | 1 | 0 | 0 | 0 | 2
Worsening speech (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 2 | 0
Albulia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 5 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 1 | 9 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 6 | 0
Euphoria (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 6 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Anosmia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 5 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Nasal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Acne on face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Blisters from herpes zoster infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Intertriginous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Redness on scalp due to Optune device (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Redness on upper back (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin irritation from Optune device (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 18 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT02311582/Prot_SAP_000.pdf